CLINICAL TRIAL: NCT05912738
Title: Preliminary Cohort Study on Muscle Elasticity Ultrasound Evaluation and Pathophysiological Changes in Postherpetic Neuralgia
Brief Title: Muscle Elasticity Assessment of Postherpetic Neuralgia Using Elasticity Ultrasound
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: UEL1
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2023-12

CONDITIONS: Shear Wave Elastography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PHN Patients (Self-Controlled Design): This cohort comprises the affected and unaffected side muscles in postherpetic neuralgia (PHN) patients. These muscles will undergo elasticity ultrasound assessment at baseline and post-treatment. Additionally, muscle biopsies will be performed at specific time points during the treatment period, including during interventional therapy, to analyze pathological changes and elucidate the treatment's pathophysiological effects on the affected muscles.
  Interventions: Other: Interventional therapy

INTERVENTIONS:
Other: Interventional therapy — Interventional therapy for postherpetic neuralgia includes nerve blocks, pulsed radiofrequency therapy, etc

SUMMARY:
Herpes zoster (HZ), also known as shingles, is caused by the varicella-zoster virus (VZV). Approximately 1/4 of the global population is affected by HZ, with statistics showing that about 90% of shingles patients experience acute neuralgia, and about 1/3 develop postherpetic neuralgia (PHN) after shingles. In PHN patients, about 30%-50% of the pain can persist for more than one year, and some cases can last for more than 10 years. PHN is a common complication of HZ characterized by intense pain in the area where the rash has healed, often described as burning, electric shock-like, or stabbing pain, severely affecting patients' sleep, emotions, work, and daily life. Additionally, approximately 43% of PHN patients exhibit symptoms of toxic anxiety or depression, significantly impacting their quality of life and increasing the societal burden. Due to the global aging population, the incidence of HZ and PHN is expected to significantly increase in the next 10 years, making effective prevention and treatment of PHN an urgent health issue. Although various treatments are available for PHN, a small number of patients remain unresponsive to multiple therapies, resulting in treatment-resistant chronic pain. The lack of a clear understanding of the underlying mechanisms contributes to the suboptimal treatment outcomes for PHN. Elastography, a technique that quantifies the mechanical properties of tissues by measuring their natural elasticity, trauma, degeneration, and healing processes, has shown promise as an innovative approach. Shear wave elastography (SWE) has been used to study the biomechanical characteristics of skeletal muscles by measuring the propagation speed of shear waves induced by ultrasound to quantify the shear elastic modulus, which characterizes the stiffness of soft tissues. In this study, the investigators intend to use elastography to observe the elasticity of muscle tissue in the lesions of PHN patients, with the unaffected side serving as a control. Elastography offers non-invasive, convenient, and straightforward advantages, further contributing to providing new directions for treatment and revealing the role of muscle tissue in PHN by offering new evidence. It also offers new treatment options and targets for PHN patients. While treatment of PHN is primarily focused on neural mechanisms due to HZ's neurotropism nature, recent evidence suggests that muscle tissues within the affected regions may also experience pathological changes, that contribute to the pain. These changes could reveal novel therapeutic targets and enhance patient prognosis. This study aims to investigate these muscular changes and explore myogenic pain mechanisms in PHN patients. It employs ultrasound elastography to compare muscle elasticity between the affected and unaffected sides and conduct muscle biopsies for pathophysiological analysis to uncover the underlying mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older, diagnosed with PHN that affects the thoracic nerves and in need of surgical intervention, have been recruited. Written informed consent was obtained from all participants before inclusion. Exclusion Criteria:
* neuromuscular diseases; ongoing use of muscle relaxants and/or other medications that impact muscles; allergy to local anesthetic; a body mass index (BMI) over 30kg/m2; malignant tumors; and pregnancy. Patients who previously had surgery in the PHN-affected area or had another disease causing muscle changes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postherpetic neuralgia patients often experience unilateral symptoms, with lesions predominantly occurring on one side of the chest wall. Shear wave elastography (SWE) has been used to study the biomechanical characteristics of skeletal muscles by measuring the propagation speed of shear waves induced by ultrasound to quantify the shear elastic modulus, which characterizes the stiffness of soft tissues. Therefore, the investigators intend to use elastography to observe the elasticity of muscle tissue in the lesions of PHN patients, with the unaffected side serving as a control.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-08-14 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Shear Wave Elastography | up to 1 month
  Shear-wave elastography has recently emerged as a promising assessment tool with the potential for diagnosing and monitoring muscle changes and as a noninvasive method to estimate muscle.

SECONDARY OUTCOMES:
A comparison of muscle elasticity between the affected and contralateral healthy sides across different PHN stages | up to 3 months
A comparison of the before and after the interventional therapy of SWE measurements | up to 3 months
A comparison SWE of measurements between groups receiving conventional treatment alone and those receiving conventional treatment plus targeted muscle relaxation therapy | up to 3 months
A comparison of the histopathological data of the muscle samples from the affected and the unaffected sides | up to 3 months
A comparison of the NRS pain scores before and after the treatment, document the number of treatment sessions, and analyze the duration of PHN | up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Xulei Cui, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking union medical college hospital, Beijing, Beijing Municipality, China